CLINICAL TRIAL: NCT05493904
Title: Impact of Optical Coherence Tomography-guided Versus Angiography-guided Stent Optimization on Post-Interventional Fractional Flow Reserve in Patients With Complex Coronary Artery Lesions
Brief Title: PREcise Percutaneous Coronary Intervention for Stent OptimizatION in Treatment of COMPLEX Lesion (PRECISION-COMPLEX)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Seung Hun Lee, Clinical Assistant Professor, Chonnam National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNUH-2022-283
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease; Angina Pectoris
Keywords: Percutaneous Coronary Intervention; Intravascular Imaging; Optical Coherence Tomography; Fractional Flow Reserve; Complex Lesion
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OCT-guided PCI arm (Active Comparator): Use of OCT will be strongly recommended at any step of PCI (pre-PCI, during PCI and post-PCI), but OCT evaluation after stent implantation will be mandatory. In case of staged procedure during the same hospitalization, following the initially allocated strategy would be strongly recommended.
  Interventions: Procedure: OCT-guided PCI; Device: Drug-eluting stent
- Angiography-guided PCI arm (Active Comparator): The PCI procedure in this group will be performed as standard procedure. After deployment of stent, stent optimization will be done based on angiographic findings. In case of staged procedure during the same hospitalization, following the initially allocated strategy would be strongly recommended.
  Interventions: Procedure: Angiography-guided PCI; Device: Drug-eluting stent

INTERVENTIONS:
Procedure: OCT-guided PCI — For patients randomly allocated to this arm, PCI for complex lesions will be performed using OCT.
  OCT Reference site: Most normal looking segment, No Lipidic plaque. Operator can decide 1 of 2 methods for stent sizing.
  1. By measuring vessel diameter at the distal reference sites (in case of ≥180° of the external elastic membrane [EEL] can be identified). In this case, stent diameter will be determined using mean external elastic membrane diameter at the distal reference, rounded down to the nearest 0.25mm (Ex> mean external elastic membrane reference diameter 3.35mm, 3.25mm stent diameter will be chosen).
  2. By measuring lumen diameter at the distal reference sites (in case of ≥180° of the external elastic membrane cannot be identified). In this case, stent diameter will be determined using mean lumen diameter at the distal reference, rounded up to the nearest 0.25mm (Ex> mean distal reference lumen diameter 2.55mm, 2.75mm stent diameter will be chosen).
  Arms: OCT-guided PCI arm
Procedure: Angiography-guided PCI — For patients randomly allocated to this arm, PCI for complex lesions will be performed using angiography only.
  The optimization guided by angiography should meet the criteria of angiographic residual diameter stenosis less than 30% by visual estimation and the absence of flow limiting dissection (≥Type C dissection). When angiographic under-expansion of the stent is suspected, adjunctive balloon dilatation will be strongly recommended.
  Arms: Angiography-guided PCI arm
Device: Drug-eluting stent — All patient will be received percutaneous coronary intervention with second generation drug-eluting stent.

SUMMARY:
The aim of the study is to compare post-interventional fractional flow reserve (FFR) value between optical coherence tomography(OCT)-guided and angiography-guided strategy for treatment of complex coronary lesion.

DETAILED DESCRIPTION:
There has been ample evidence of the role of intracoronary imaging for optimizing the stent, especially among the patients with complex coronary lesions. Intracoronary imaging can be used during the entire process of percutaneous coronary intervention (PCI), from pre-PCI to post-PCI stages. Notably, approximately 15-20% of patients who underwent angiographically successful PCI showed significant stent underexpansion, malapposition, intra-stent thrombus formation, and edge dissection on intracoronary imaging studies, including optical coherence tomography (OCT).

Meanwhile, the role of pre-interventional fractional flow reserve (FFR) measurement has been well established and recommended by recent guideline. However, although previous studies evaluated the efficacy and safety of FFR-guided decision-making followed by angiographic stent implantation, they did not evaluate functionally optimized revascularization. Actually, the vessels with low post-PCI FFR had substantial proportions of suboptimized stented (underexpansion and acute malapposition) and residual disease in non-stented segments. Furthermore, several large observational studies have suggested that suboptimal physiologic results after PCI is associated with an increased risk of clinical events. Previously, the DOCTORS trial found out that OCT-guided PCI was associated with higher post-PCI FFR than angiography-guided PCI (0.94±0.04 vs. 0.92±0.05, P=0.005).

Therefore, OCT can be a useful tool for acquiring functional optimal results after stent implantation. This synergic effect between OCT and post-PCI FFR can be maximized when the investigators perform PCI for complex lesions. This study sought to evaluate compare post-interventional FFR value between OCT-guided and angiography-guided strategy for treatment of complex coronary lesion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years old
2. Patients with stable or unstable angina and complex coronary lesions*
3. Patients who were indicated revascularization

   * Diameter stenosis >90% by angiography
   * Diameter stenosis with 50~90% with pre-interventional FFR ≤0.80
4. Patients who underwent implantation of 2nd generation drug-eluting stent

   * Definitions of complex coronary lesions

     1. True bifurcation lesion (Medina 1,1,1/1,0,1/0,1,1) with side branch ≥2.5mm size
     2. Chronic total occlusion (≥3 months) as target lesion
     3. PCI for unprotected left main (LM) disease (LM os, body, distal LM bifurcation including non-true bifurcation)
     4. Long coronary lesions (implanted stent ≥38 mm in length)
     5. Multi-vessel PCI (≥2 major epicardial coronary arteries treated at one PCI session)
     6. Multiple stents needed (≥3 more stent per patient)
     7. In-stent restenosis lesion as target lesion
     8. Severely calcified lesion (encircling calcium in angiography)
     9. Left anterior descending (LAD), left circumflex artery (LCX), and right coronary artery (RCA) ostial lesion

Exclusion Criteria:

1. Target lesions not amenable for PCI by operators' decision
2. Cardiogenic shock (Killip class IV) at presentation
3. Less than TIMI 3 flow of target vessel after index procedure
4. Intolerance to Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Heparin, Everolimus, Zotarolimus, Biolimus, or Sirolimus
5. Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)
6. Renal insufficiency such that an additional contrast medium would be harmful for patient
7. Recent ST-segment elevation myocardial infarction (STEMI)
8. Inability to receive adenosine or nicorandil injection
9. Pregnancy or breast feeding
10. Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment)
11. Unwillingness or inability to comply with the procedures described in this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Suboptimal post-PCI physiological results | Immediate after the index procedure
  Proportion of patients with a final post-interventional fractional flow reserve <0.85

SECONDARY OUTCOMES:
Rate of target vessel failure (TVF) | 2 years after last patient enrollment
  a composite of cardiac death, target-vessel myocardial infarction (MI), and target-vessel revascularization (TVR)
Rate of all-cause death | 2 years after last patient enrollment
  death from any-cause
Rate of cardiac death | 2 years after last patient enrollment
  death from cardiac-cause
Rate of target vessel MI without periprocedural MI | 2 years after last patient enrollment
  Myocardial infarction without periprocedural myocardial infarction
Rate of target vessel MI with periprocedural MI | 2 years after last patient enrollment
  Myocardial infarction with periprocedural myocardial infarction
Rate of target lesion revascularization (TLR) | 2 years after last patient enrollment
  ischemia-driven or all
Rate of target vessel revascularization (TVR) | 2 years after last patient enrollment
  ischemia-driven or all
Rate of any MI | 2 years after last patient enrollment
  any myocardial infarction
Rate of any revascularization | 2 years after last patient enrollment
  ischemia-driven or all
Rate of stent thrombosis | 2 years after last patient enrollment
  definite, probable, or possible
FFR gain between pre- and post-interventional stages | Immediate after the index procedure
  [Post-interventional fractional flow reserve value] - [Pre-interventional fractional flow reserve value]
Trans-stent FFR gradient | Immediate after the index procedure
  FFR gradient across the stent (ΔFFRstent)
Post-interventional non-hyperemic pressure ratios | Immediate after the index procedure
  Values of post-PCI non-hyperemic pressure ratios

OTHER OUTCOMES:
Incidence of contrast-induced nephropathy | 48-72 hours after index procedure
  defined as an increase in serum creatinine of ≥0.5mg/dL or ≥25% from baseline after contrast agent exposure
Total procedure time | Immediate after the index procedure
  Total procedure time
Total amount of contrast dose | Immediate after the index procedure
  Total amount of contrast dose
Total fluoroscopy time | Immediate after the index procedure
  Total fluoroscopy time
Total amount of radiation dose | Immediate after the index procedure
  Total amount of radiation dose

CONTACTS AND LOCATIONS:
Overall Officials: Youngkeun Ahn, MD, PhD, Study Chair — Chonnam National University Hospital
Locations (4):
- South Korea (4):
  - Chonnam National University Hospital, Gwangju
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after study completion
Access Criteria: After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT05493904/Prot_SAP_003.pdf